CLINICAL TRIAL: NCT01232231
Title: Comprehensive Strategy to Decolonize Methicillin-resistant Staphylococcus Aureus in the Outpatient Setting: a Randomized Controlled Study
Brief Title: Comprehensive Strategy to Decolonize Methicillin-resistant Staphylococcus Aureus (MRSA) in the Outpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Kim (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor-Investigator, Joseph Kim, Clinical Assistant Professor, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E23134
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Methicillin-resistant Staphylococcus Aureus
Keywords: methicillin-resistant Staphylococcus aureus; decolonization; random allocation; outpatient
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- decolonization treatment (Active Comparator): topical antiseptic, intranasal antimicrobial, and oral antimicrobial that have activity against MRSA in addition to education regarding personal hygiene and environmental cleaning
  Interventions: Drug: pharmacological decolonization treatment
- education (Other): No decolonization treatment in addition to education regarding personal hygiene and environmental cleaning
  Interventions: Behavioral: Education

INTERVENTIONS:
Drug: pharmacological decolonization treatment — Chlorhexidine gluconate 4% body scrub and 2% shampoo daily PLUS mupirocin 2%, fusidic acid 2%, or chlorhexidine gluconate 0.2% intranasally bid PLUS trimethoprim-sulfamethoxazole 160/800mg po bid or doxycycline 100mg po bid all for 7 days
  Arms: decolonization treatment
Behavioral: Education — No pharmacological decolonization treatment but given education regarding personal hygiene and environmental cleaning
  Arms: education

SUMMARY:
The purpose of this study is to determine the effectiveness of topical and oral antibiotics in eliminating carriage of methicillin-resistant Staphylococcus aureus (MRSA) among those living in the community. We hypothesize that a greater proportion of those who receive intervention will eliminate MRSA carriage compared to those who do not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Prior MRSA infection (i.e index case)
* Identified as being colonized with MRSA on initial screen

Exclusion Criteria:

* Are pregnant or breastfeeding.
* Have indwelling catheters.
* Received prior decolonization treatment within last 6 months of enrollment.
* Have allergy to study medication.
* Are colonized with MRSA strain resistant to study medication.
* Have active infection requiring systemic antimicrobials.
* Are household contacts to index case.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Eradication of MRSA carriage | 90 days after randomization

SECONDARY OUTCOMES:
Occurrence of MRSA infection | Within 6 months of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Louie, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada